CLINICAL TRIAL: NCT06808724
Title: Clinical Influence of Different Surface Treatments on Implant Stabiity: a Prospective Observational Clinical Study
Brief Title: Clinical Influence of Different Surface Treatments on Implant Stabiity
Status: Recruiting | Type: Observational
Sponsor: International Piezosurgery Academy (Other)
Collaborators: University of Trieste (Other)
Responsible Party: Sponsor
Other Study IDs: IMPLANT SURFACE MODIFICATIONS
Record Dates: First submitted 2025-01-21; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Edentulous Alveolar Ridge
MeSH Terms: interventions — Drug Implants

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Test: ozonated oil / plasma activation
  Interventions: Procedure: implant with ozonated oil; Procedure: implant with plasma activation
- Control: No surface treatment
  Interventions: Procedure: non-activated implant

INTERVENTIONS:
Procedure: implant with ozonated oil — Following local anesthesia (mepivacaine HCl 2% with epinephrine 1:100,000), a minimally invasive full-thickness flap will be elevated. Implant site preparation will be performed with twist drills. Ozonated oil (Surgy O3) will be applied to the implant surface and then the implant will be inserted into the prepared osteotomy site. A 3 mm high transepithelial abutment will be then screwed using a torque wrench, tightened to 30 Ncm. Single monofilament synthetic polypropylene 4.0 sutures will be used to close the flaps.
  Groups: Test
Procedure: non-activated implant — Following local anesthesia (mepivacaine HCl 2% with epinephrine 1:100,000), a minimally invasive full-thickness flap will be elevated. Implant site preparation will be performed with twist drills. In the control group, the implant will be inserted without any treatment. A 3 mm high transepithelial abutment will be then attached using a torque wrench, tightened to 30 Ncm. Single monofilament synthetic polypropylene 4.0 sutures will be used to close the flaps.
  Groups: Control
Procedure: implant with plasma activation — Following local anesthesia (mepivacaine HCl 2% with epinephrine 1:100,000), a minimally invasive full-thickness flap will be elevated. Implant site preparation will be performed with twist drills. Implant will undergo vacuum-plasma activation immediately before insertion (Plasma X Motion, Megagen, Gyeongbuk, South Korea) and then it will be inserted into the prepared osteotomy site. A transepithelial abutment will then be attached using a torque wrench, tightened to 30 Ncm. Single monofilament synthetic polypropylene 4.0 sutures will be used to close the flaps.
  Groups: Test

SUMMARY:
The goal of this observational study is to monitor, within a cohort of patients requiring rehabilitation at two different sites in the premolar area, the primary and secondary stability of implants placed with different surface treatments: vacuum-plasma activation, ozonated oil and non-activated implants.

DETAILED DESCRIPTION:
The primary outcome measures included primary implant stability, assessed through insertion torque and the Implant Stability Quotient (ISQ).

Secondary outcome measures included the pattern of implant secondary stability during the first 90 days post-implant placement (ISQ), implant survival after one year, NPRS comparison between treatments at one week postoperatively, and any complications or adverse events.

As an additional objective, the study aimed to assess whether a relationship existed between implant surface treatment and early marginal bone loss. Marginal bone levels were measured at three time points: immediately after surgery (T0), upon delivery of prosthetic rehabilitation (T1), and after one year of loading (T2). The distance between the implant platform and the bone crest was measured at each interval, on both the mesial and distal aspects of the implant. A positive value was assigned when the bone crest was coronal to the implant platform, whereas a negative value was assigned when the bone crest was apical to the implant platform.

Study Design: Observational, prospective, non-profit case-control study.

Study Population: The study will be conducted in an outpatient hospital setting.

Enrollment Procedure: All patients meeting the inclusion and exclusion criteria will be enrolled in the study after receiving the Information Sheet and providing written informed consent.

Patients seeking implant-supported rehabilitation due to the absence of at least two teeth were initially evaluated with a periapical radiograph of the selected sites to assess residual bone height adequacy. If sufficient bone height was observed, a second-level radiographic examination using Cone Beam Computed Tomography (CBCT) was performed to confirm the adequacy of bone volume for implant rehabilitation.

Surgical Phase: Following local anesthesia (mepivacaine HCl 2% with epinephrine 1:100,000), a minimally invasive full-thickness flap was elevated. The same surgeon performed all procedures. Implant site preparation was performed using twist drills. In one group, ozonated oil (Surgy O3, Biosanity) was applied to the implant surface and then the implant was inserted into the prepared osteotomy site. A transepithelial abutment was then attached using a torque wrench, tightened to 30 Ncm. In the second group, implant underwent vacuum-plasma activation immediately before insertion (Plasma X Motion, Megagen, Gyeongbuk, South Korea) and then it was inserted into the prepared osteotomy site. A transepithelial abutment was then attached using a torque wrench, tightened to 30 Ncm. In the control group, the implant was inserted without any treatment. A transepithelial abutment was then attached using a torque wrench, tightened to 30 Ncm. Single monofilament synthetic polypropylene 4.0 sutures were used to close the flaps.

A postoperative radiographic assessment was conducted to verify correct implant positioning.

A blinded operator measured ISQ values for each implant in two directions: vestibular-palatal and mesio-distal. Measurements were taken at the abutment level three times per direction, and the averages were used for statistical analysis.

ISQ measurements were performed using a Resonance Frequency Analysis (RFA) device (Osstell, Göteborg, Sweden) with the appropriate transducer for the selected abutment (Smartpeg Type 05, Osstell, Göteborg, Sweden).

Follow-up: After surgery, a follow-up visit was scheduled after one week for suture removal, soft tissue healing assessment, and ISQ measurements. Additional follow-ups occurred at 14, 21, 28, 42, 56, and 90 days, with the same parameters reassessed at each visit.

All implants were restored with screw-retained single metal-ceramic crowns four months after surgery and were followed up for at least 12 months after prosthetic loading. Radiographic check-ups were conducted at 6 months and 1 year.

For the sample size calculation, it was assumed that the minimal clinically relevant difference between the groups was 5 points on the ISQ scale, with a standard deviation of 5. Using an 80% power and a 95% significance level, the calculation yielded a sample size of approximately 16 participants per group (rounded to the next whole number). This ensures sufficient power to detect the anticipated difference between the groups.

Statistical Plan: Statistical analysis will be performed using a computerized statistical package (SigmaStat 3.5, SPSS Inc., Germany). Data will be expressed as mean ± standard deviation or median (interquartile range) for parametric and non-parametric values, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Age older than 18 years old;
* Indication for an implant-supported rehabilitation in the left and right upper premolar/first molar areas;
* The area in which the implants will be placed must have had at least 6 months of healing;
* No use of grafts or bone substitutes following tooth extraction;
* Bone volume measuring at least 10 mm in height and 6 mm in width;
* Absence or decision to not wear a removable prosthesis during the healing period;
* Patients with good and stable oral hygiene;
* Signed informed consent form.

Exclusion Criteria:

* Acute myocardial infarction within the previous six months;
* Uncontrolled bleeding disorders;
* Uncontrolled diabetes (HBA1c > 7.5%);
* Radiotherapy in the head-neck area in the previous 48 months;
* Immunocompromised patients (es. AIDS / chemotherapy);
* Current or previous treatment with antiresorptive drugs via intravenous injection;
* Psychological or psychiatric disease;
* Alcohol and /or drugs abuse;
* Heavy smokers (more than 10 cigarettes / day);
* Plaque index >20% and/or bleeding on probing >10%
* Pregnant or breastfeeding patients;
* Patients refusing to participate in follow-up checks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: After investigating general and local anamnesis, which included evaluation of systemic illnesses and potential allergies, a dental visit was conducted to formulate a specific treatment plan.
  If the patient was deemed eligible for the research protocol, an additional periapical radiograph was obtained for each selected site to assess the adequacy of residual bone height.
  If the available bone height appeared to be sufficient, a second-level radiographic exam, a Cone Beam Computed Tomography (CBCT), was performed to evaluate whether the bone volume was adequate for supporting implant rehabilitation.
  For patients requiring tooth extraction, this second assessment was performed after six months of healing after extraction.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2025-01-31 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Implant primary stability measured with RFA device (Osstell) | Immediately after implant placement
  Resonance Frequency Analysis (RFA) device (Osstell, Göteborg, Sweden) with the appropriate transducer for the selected abutment (Smartpeg Type 05, Osstell, Göteborg, Sweden)
Implant primary stability in Newton | Immediately after implant placement
  Insertion torque

SECONDARY OUTCOMES:
Implant secondary stability measured with RFA device (Osstell) | 7 days after implant insertion
  Resonance Frequency Analysis (RFA) device (Osstell, Göteborg, Sweden) with the appropriate transducer for the selected abutment (Smartpeg Type 05, Osstell, Göteborg, Sweden)
Implant secondary stability measured with RFA device (Osstell) | 14 days after implant insertion
  Resonance Frequency Analysis (RFA) device (Osstell, Göteborg, Sweden) with the appropriate transducer for the selected abutment (Smartpeg Type 05, Osstell, Göteborg, Sweden)
Implant secondary stability measured with RFA device (Osstell) | 21 days after implant insertion
  Resonance Frequency Analysis (RFA) device (Osstell, Göteborg, Sweden) with the appropriate transducer for the selected abutment (Smartpeg Type 05, Osstell, Göteborg, Sweden)
Implant secondary stability measured with RFA device (Osstell) | 28 days after implant insertion
  Resonance Frequency Analysis (RFA) device (Osstell, Göteborg, Sweden) with the appropriate transducer for the selected abutment (Smartpeg Type 05, Osstell, Göteborg, Sweden)
Implant secondary stability measured with RFA device (Osstell) | 42 days after implant insertion
  Resonance Frequency Analysis (RFA) device (Osstell, Göteborg, Sweden) with the appropriate transducer for the selected abutment (Smartpeg Type 05, Osstell, Göteborg, Sweden)
Implant secondary stability measured with RFA device (Osstell) | 56 days after implant insertion
  Resonance Frequency Analysis (RFA) device (Osstell, Göteborg, Sweden) with the appropriate transducer for the selected abutment (Smartpeg Type 05, Osstell, Göteborg, Sweden)
Implant secondary stability measured with RFA device (Osstell) | 90 days after implant insertion
  Resonance Frequency Analysis (RFA) device (Osstell, Göteborg, Sweden) with the appropriate transducer for the selected abutment (Smartpeg Type 05, Osstell, Göteborg, Sweden)

OTHER OUTCOMES:
Peri-implant marginal bone level stability | Immediately after surgery
  The distance between implant platform and bone crest was measured at each time interval, on both mesial and distal aspects of the implant. A positive value was assigned when the bone crest was coronal to the implant platform, whereas a negative value was assigned when the bone crest was apical to the implant platform.
  MBL has no defined minimum or maximum value.
Peri-implant marginal bone level stability | Upon delivery of prosthetic rehabilitation (6 months after surgery)
  The distance between implant platform and bone crest was measured at each time interval, on both mesial and distal aspects of the implant. A positive value was assigned when the bone crest was coronal to the implant platform, whereas a negative value was assigned when the bone crest was apical to the implant platform.
  MBL has no defined minimum or maximum value.
Peri-implant marginal bone level stability | One year of loading
  The distance between implant platform and bone crest was measured at each time interval, on both mesial and distal aspects of the implant. A positive value was assigned when the bone crest was coronal to the implant platform, whereas a negative value was assigned when the bone crest was apical to the implant platform. MBL has no defined minimum or maximum value.
NPRS | 7 days after implant insertion
  Numeric Pain Rating Scale between the treatments (minimum 0, maximum 10)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Trieste, Trieste, TS, Italy

IPD SHARING:
Plan to Share IPD: No